CLINICAL TRIAL: NCT05149937
Title: Development and Testing of an Interprofessional, Person-centered Care Concept for People Living at Home With Care Needs.
Acronym: interprof HOME
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped before first patient inclusion.
  Mixed-methods-study (part a) completed per protocol, explorative survey (part b) withdrawn due to organizational reasons
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Karsten Gavenis, Clinical Study Management on behalf of the Principal Investigator, University Medical Center Goettingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-00425
Record Dates: First submitted 2021-11-03; First posted 2021-12-08 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Utilization of Nursing, Medical and Therapeutical Care of People Living at Home With Care Needs
Keywords: interprofessional collaboration; reduction of hospitalisation; people living at home with care needs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional group (Experimental): Implementation of interprof Home measures to improve cooperation between nursing services, general practitioners and members of the therapeutic professions in the care of people living at home with care needs.
  Interventions: Other: interprofessional, person-centered care concept

INTERVENTIONS:
Other: interprofessional, person-centered care concept — interprofessional, person-centered care concept

SUMMARY:
The aim of the project is to develop and pilot measures to optimize the person-centered cooperation between nursing services, general practitioners and members of the therapeutic professions in the care of people living at home with care needs, so that hospital admissions and the use of unplanned medical and rescue services are avoided, the quality of life is improved and a deterioration in the need for long-term care can be stopped.

This is done by developing an interprofessional person-centered collaboration-concept, perform an explorative mixed-methods-study: interviews, focus groups, expert workshops, survey of best practices, shadowing, questionnaires.

DETAILED DESCRIPTION:
Description of mixed-methods-study:

1. Interviews with

   * 20 patients,
   * 20 relatives,
   * 5 experts of health insurance professionals,
   * and 3 focus groups à 8 persons with general practioniers, nurses, therapists.
2. investigation of best practice cases
3. explorative survey of 100 cases in each group:

   * general practitioner
   * nursing services
   * therapists
   * persons in need of care
   * family members of persons in need of care

The mixed-methods-study is analysed in different ways:

* structured content analysis
* case-based qualitative analysis of interviews
* descriptive analysis

The mixed-methods-study has been approved by the ethics committee and is recruiting.

ELIGIBILITY:
Inclusion Criteria:

* years of age >18
* receipt of benefits in the form of outpatient care according to SGB XI,
* preliminary / final classification of care ≥level 2
* expected life expectancy >6 months
* informed consent
* sufficient opportunity to answer answering questions about patient-reported outcomes

Exclusion Criteria:

* Living in nursing home / planned move-in within the following 6 months
* claim acceptance of SAPV
* participation in scientific study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
cumulative number of hospitalisation | 40 months
  Cumulative incidence of hospitalisations within 12 months

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tetzlaff B, Mazur AL, Sekanina U, Huckle T, Dano R, Hockelmann C, Diel M, Bremer L, Kuhn A, Romanski AM, Kuba S, Ruppel T, Balzer K, Kopke S, Maurer I, Weber CE, Scherer M, Hummers E, Muller CA. Development of an interprofessional person-centred care concept for persons with care needs living in their own homes in Germany (interprof HOME): a mixed methods study. BMC Prim Care. 2025 Nov 15;26(1):363. doi: 10.1186/s12875-025-03098-0. PMID 41241758
- [Derived] Sekanina U, Tetzlaff B, Mazur A, Huckle T, Kuhn A, Dano R, Hockelmann C, Scherer M, Balzer K, Kopke S, Hummers E, Muller C. Interprofessional collaboration in the home care setting: perspectives of people receiving home care, relatives, nurses, general practitioners, and therapists-results of a qualitative analysis. BMC Prim Care. 2024 Mar 4;25(1):79. doi: 10.1186/s12875-024-02313-8. PMID 38438843
- [Derived] Tetzlaff B, Scherer M, Balzer K, Steyer L, Kopke S, Friede T, Maurer I, Weber CE, Konig HH, Konnopka A, Ruppel T, Mazur A, Hummers E, Mueller CA. Development of an interprofessional person-centred care concept for persons with care needs living in their own homes (interprof HOME): study protocol for a mixed-methods study. BMJ Open. 2023 Jul 14;13(7):e069597. doi: 10.1136/bmjopen-2022-069597. PMID 37451715